CLINICAL TRIAL: NCT05575479
Title: Physical Activity Behavior and Health-Related Quality of Life in Parkinson's Disease Patients: Role of Social Cognitive Variables
Brief Title: PA Behavior and HRQoL in Parkinson's Disease Patients Patients: Role of Social Cognitive Variables
Acronym: PDQ
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Brian Focht, Associate Professor of Kinesiology Department of Human Sciences, Ohio State University
Other Study IDs: 2015B0259
Record Dates: First submitted 2015-09-14; First posted 2022-10-12 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Parkinson Disease; Idiopathic Parkinson Disease; Idiopathic Parkinson's Disease; Parkinson Disease, Idiopathic; Parkinson's Disease; Parkinson's Disease, Idiopathic
Keywords: Social Cognitive Theory; Physical Activity; Quality of Life; Parkinsons
MeSH Terms: conditions — Parkinson Disease; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Idiopathic Parkinson's Patients: Patients with idiopathic parkinson's disease

SUMMARY:
The primary aim of the study will be to examine Social Cognitive Theory (SCT) correlates, of physical activity (PA) participation and health-related quality of life (HRQoL) in Parkinson's disease participants.

DETAILED DESCRIPTION:
The body of evidence in the physical therapy and rehabilitation literature supports that physical activity is associated with improvements in quality of life for Parkinson's Disease (PD) patients. However, few studies have examined the underlying variables that may account for this relationship in PD patients. Researchers have examined stages of readiness to exercise in PD patients and barriers to exercise and found a strong association between self-efficacy and exercise in PD patients, rather than disability .

Researchers suggest that social cognitive theory (SCT) constructs are important correlates of physical activity for PD patients and should be targeted in interventions. A more comprehensive study of SCT correlates - Self-Efficacy (SE), Outcome Expectations (OE), and Self-Regulation (SR) should provide a better understanding of the factors that contribute to physical activity participation and the physical activity / health-related quality of life relationship in PD patients.

ELIGIBILITY:
Inclusion Criteria:

1. English speaking
2. Parkinson's disease diagnosed by a neurologist

Exclusion Criteria:

1. Atypical Parkinson's
2. Supranuclear Palsy
3. Deep Brain Stimulation (DBS) or other brain surgery
4. Not living independently (living in assisted-living or skilled-nursing facility)
5. Spouse or caregiver responding instead of PD participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators are using a cross-sectional experimental design of 404 geographically diverse Parkinson's participants. Physiologic (Hoehn & Yahr) and psychological (surveys and single-item measures) measures will be collected via web-based surveys in Qualtrics accessed through a link.
  Sample Using (Fritz & MacKinnon, 2007) article on the required sample size necessary to detect mediated effects, using the empirical estimates in Table 3 for the Baron and Kenny test with ť = .59, α = .59 and β = .14, the desired sample size needed for a power of .8 would be 404. In this population, the investigators expect that some PD participants may start the survey and be unable to finish. For this reason, the investigators would like to oversample by 25% with a target of 505 participants.
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2015-08; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Health-Related Quality of Life (HRQoL) correlation to self-reported physical activity (PA) | participant's respond to survey questions only 1 time
  multiple linear regression analysis will be used to determine if higher HRQoL is significantly related to self-reported physical activity in PD patients.

SECONDARY OUTCOMES:
Self-efficacy (SE), Outcomes Expectations (OE), and Self-Regulation (SR) correlation to self-reported HRQoL | Outcomes as measured at a single baseline assessment
  multiple linear regression analysis will be used to determine if higher levels of SE, OE, and SR are significantly related to self-reported HRQoL.

OTHER OUTCOMES:
Social Cognitive Theory (SCT) constructs as mediators between self-reported PA and HRQoL | Outcomes as measured at a single baseline assessment
  hierarchical linear regression model will be used to examine the SCT constructs as potential mediators between self-reported PA and HRQoL in PD patients. Also, any variables determined to have significant impact in the multiple regression models will be controlled for in the HLM, allowing us to investigate the effects of certain variables while controlling for the effects of others.
SCT constructs correlation to self-reported PA | Outcomes as measured at a single baseline assessment
  multiple linear regression analysis will then be used to examine the relationship between the social cognitive theory constructs and self-reported physical activity in PD patients.

CONTACTS AND LOCATIONS:
Overall Officials: Brian C Focht, PhD, Principal Investigator — Associate Professor Kinesiology
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

REFERENCES:
- See also: Qualtrics Survey Study Link — http://tinyurl.com/p5h58to